CLINICAL TRIAL: NCT02544932
Title: Prospective Randomized Study for Evaluating Vascular Protective Effects of New Oral Anticoagulants in High Risk Patients With Atrial Fibrillation
Brief Title: Pleotropic Effect of New Oral Anticoagulants
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Weon Kim, professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREFER-AF
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Atrial Fibrillation
Keywords: anticoagulant; atherosclerosis; endothelium
MeSH Terms: conditions — Atrial Fibrillation; Atherosclerosis | interventions — Dabigatran; Rivaroxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- dabigatran 110mg or 150mg (Experimental): After once enrolled, subjects will be randomized to dabigatran group. (110mg or 150mg twice a day)
  Interventions: Drug: dabigatran
- ribaroxaban 20mg (Experimental): After once enrolled, subjects will be randomized to ribaroxaban group. (20mg once daily)
  Interventions: Drug: ribaroxaban
- warfarin (Active Comparator): After once enrolled, subjects will be randomized to warfarin group. (controlled by INR 2-3)
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: dabigatran — After randomization, patients of this group was will be treated to dabigatran 110mg or 150mg twice a day for 24months
  Other Names: pradaxa
  Arms: dabigatran 110mg or 150mg
Drug: ribaroxaban — After randomization, patients of this group was will be treated to ribaroxaban 20mg once a day for 24months.
  Other Names: xarelto
  Arms: ribaroxaban 20mg
Drug: Warfarin — After randomization, patients of this group was will be treated to warfarin and controlled by INR 2-3 for 24months.
  Arms: warfarin

SUMMARY:
Atrial fibrillation (AF) has been known to have several pathophysiologic mechanisms including endothelial dysfunction of heart and vessel. This study was designed to determine the efficacy of NOAC therapy in the prevention of endothelial dysfunction and progression of atherosclerosis of AF subjects.

DETAILED DESCRIPTION:
The properties of oral, direct inhibitors of factor Xa (e.g. rivaroxaban) and thrombin (e.g. dabigatran) have been examined the haemostasis and thromboembolism management. Preclinical studies have provided evidences for the effects of direct factor Xa or thrombin inhibition beyond anticoagulation, including anti-inflammatory and protective activities in atherosclerotic plaque development . Therefore, this study evaluates the protective effects of NAOC with the reactive hyperemia peripheral arterial tonometry (RH-PAT) measurements reflecting endothelial function by Endo-PAT2000 and intima-media thickness (IMT) of the carotid artery, which is used as a surrogate endpoint of atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* CHA2DS2-VASc score above 2

Exclusion Criteria:

* severe peripheral arterial disease (greater than a Fontaine IIb category)
* grade 4 or higher cerebral infarction on the Modified Rankin Scale
* proven coronary artery disease by coronary angiogram
* severe hepatic or renal dysfunction
* uncontrolled congestive heart failure
* uncontrolled hypertension or diabetes mellitus
* hematologic disorders
* allergy or hypersensitivity to the investigational drugs
* pregnant or lactating women or women wishing to become pregnant

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
The changes in reactive hyperemia index (RHI) | 12months

SECONDARY OUTCOMES:
right and left maximum IMT of the common carotid artery (CCA) | 24months
right and left mean IMT of the common carotid artery (CCA) | 24months
adverse events | 24months

CONTACTS AND LOCATIONS:
Overall Officials: Weon Kim, MD, PhD, Principal Investigator — Kyunghee University Medical Center
Locations (1):
- Kyung Hee University, Seoul, South Korea

REFERENCES:
- [Derived] Kim JB, Joung HJ, Lee JM, Woo JS, Kim WS, Kim KS, Lee KH, Kim W. Evaluation of the vascular protective effects of new oral anticoagulants in high-risk patients with atrial fibrillation (PREFER-AF): study protocol for a randomized controlled trial. Trials. 2016 Aug 24;17(1):422. doi: 10.1186/s13063-016-1541-8. PMID 27558002